CLINICAL TRIAL: NCT00182663
Title: Maintenance Therapy With Thalidomide, Dexamethasone and Clarithromycin (Biaxin) Following Autologous/Syngeneic Transplant for Multiple Myeloma
Brief Title: Thalidomide, Dexamethasone, and Clarithromycin in Treating Patients With Multiple Myeloma Previously Treated With Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1767.00; NCI-2011-00387 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-04

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Clarithromycin; Thalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (immunomodulator, antiangiogenesis, steroid therapy) (Experimental): Patients receive thalidomide PO QD dexamethasone PO once weekly, and clarithromycin PO BID. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Treatment with thalidomide continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: clarithromycin; Drug: thalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: clarithromycin — Given PO
  Other Names: Abbott-56268; Biaxin; CLARITH
Drug: thalidomide — Given PO
  Other Names: Kevadon; Synovir; THAL; Thalomid
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM

SUMMARY:
This phase II trial studies the side effects and how well giving thalidomide, dexamethasone, and clarithromycin together works in treating patients with multiple myeloma previously treated with transplant. Biological therapies, such as thalidomide and clarithromycin, may stimulate the immune system in different ways and stop cancer cells from growing. Dexamethasone also works in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving thalidomide together with dexamethasone and clarithromycin after a transplant may be an effective treatment for multiple myeloma

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the toxicity of the use of Thalidomide/Biaxin (Clarithromycin)/Dexamethasone as maintenance therapy after autologous/syngeneic transplant.

II. Evaluate the median time to disease progression. III. Evaluate survival.

OUTLINE:

Patients receive thalidomide orally (PO) once daily (QD), dexamethasone PO once weekly, and clarithromycin PO twice daily (BID). Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Treatment with thalidomide continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Any autologous or syngeneic patient who underwent high dose melphalan (>= 140 mg/m^2) therapy/peripheral blood stem cell (PBSC) or bone marrow (BM) rescue for any stage of multiple myeloma and did not participate in another clinical transplant trial which is also evaluating disease free survival or survival
* Platelet count (transfusion independent) > 50,000 cells/mm^3 for 5 calendar days after recovery from high dose
* Absolute granulocyte count > 1500 cells/mm^3 for 5 calendar days after recovery from high dose
* Patients will start therapy between 30 days to 120 days after transplant
* Willingness and ability to comply with Food and Drug Administration (FDA)-mandated S.T.E.P.S. (Celgene System for Thalidomide Education and Prescribing Safety) Program
* Signing a written informed consent form

Exclusion Criteria:

* Karnofsky score less than 70
* A left ventricular ejection fraction less than 45%; patients with congestive heart disease, history of myocardial infarction (MI), or coronary artery disease
* Total bilirubin greater than 2 mg/ml (unless history of Gilbert's disease)
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) > 2.5 x upper limit of normal
* History of deep venous thrombus, arterial occlusions, or pulmonary emboli
* Pregnant and/or lactating females
* Patients who cannot give informed consent
* Patients with untreated systemic infection
* Patients with history prior to transplant of treatment with combination therapy Thalidomide/Biaxin and Steroid without response
* Patients allergic to Thalidomide, Biaxin or Dexamethasone
* Referring physician not registered with S.T.E.P.S. program or unwilling to oversee the care of the patients on study and comply with the FDA-mandated S.T.E.P.S. Program
* Patients unwilling to practice adequate forms of contraception if clinically indicated; male patients on study need to be consulted to use latex condoms even if they have had a vasectomy every time they have sex with a woman who is able to have children while they are being treated and for four weeks after stopping drugs
* Patients with history of seizures

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-06; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Toxicity of proposed treatment with clarithromycin, dexamethasone, and thalidomide | First 3 months of therapy

SECONDARY OUTCOMES:
Time to disease progression | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States